CLINICAL TRIAL: NCT02585804
Title: Treating to Reduce Albuminuria and Normalize Hemodynamic Function in Focal ScLerosis With dApagliflozin Trial Effects: "The TRANSLATE Study"
Brief Title: Treating to Reduce Albuminuria and Normalize Hemodynamic Function in Focal ScLerosis With dApagliflozin Trial Effects
Acronym: TRANSLATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry); University of Toronto (Other); Toronto General Hospital (Other)
Responsible Party: Principal Investigator, David Z.I. Cherney, Associate Professor of Medicine, Clinician Scientist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB# 14-8284-B
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: FSGS, SGLT2, chronic kidney disease, GFR, proteinuria
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Renal Insufficiency, Chronic; Proteinuria | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapagliflozin (trade name Farxiga®) (Experimental): Oral tablet, 10mg, PO, 8 weeks
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Oral tablet, 10mg, PO, 8 weeks
  Other Names: Trade name Farxiga®

SUMMARY:
Patients with Focal Segmental Glomerulosclerosis (FSGS) constitute an increasing proportion of the total glomerulonephritis (GN) patient cohort in North America while FSGS is a risk factor for end stage renal failure. Current non-immunological FSGS therapies include the use of angiotensin converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB), to reduce intraglomerular hypertension. Unfortunately, these agents lead to incomplete renal protection. The aim of the current study is to determine whether the addition of novel sodium glucose cotransport-2 inhibitors (SGLT2i) to standard of care leads to reduced intraglomerular pressure and suppression of proteinuria. We hypothesize that combination therapy of SGLT2i drugs and conventional RAASi results in additive renal protective effects in FSGS patients. A further goal is to examine mechanisms of SGLT2 inhibition by measuring renal hemodynamic function and sodium handling. Kidney function will be assessed in FSGS patients before and after an 8 week treatment with SGLT2i dapagliflozin.

DETAILED DESCRIPTION:
FSGS and diabetic nephropathy may have common pathogenic mechanisms, that are mediated by intraglomerular hypertension, leading to hyperfiltration and proteinuria. Given that SGLT2i corrects early hemodynamic abnormalities in patients with diabetes, our aim is to determine if a similar benefit may extend to patients with FSGS. Based on previous experimental and clinical data, we hypothesize that SGLT2i will improve renal hemodynamic abnormalities characteristic of FSGS that promote renal injury and proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects diagnosed with FSGS ≥1 month prior to informed consent
* eGFR≥45 ml/min/1.73m2
* Age 18 years or greater
* No history of diabetes
* Body Mass Index (BMI) 18.5 - 45.0 kg/ m2
* Blood pressure ≥ 100/60 at screening
* Stable therapy with either an ACEi or angiotensin II receptor blocker or direct renin inhibitor for > 1 month
* >30 mg/day and <6 g/day of proteinuria unless the patient is not a candidate for immunosuppressive therapy

Exclusion Criteria:

* Leukocyte and/or nitrite positive urinalysis that is untreated;
* History of organ transplantation, cancer, liver disease;
* Bariatric surgery or other gastrointestinal surgeries that induce chronic malabsorption within the past two years;
* Current treatment with systemic corticosteroids, calcineurin inhibitors, or other immunosuppressant medications;
* Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells;
* Pre-menopausal women who are nursing, pregnant, or of child-bearing potential and not practising an acceptable method of birth control;
* Participation in another therapeutic trial with an investigational drug within 30 days prior to informed consent;
* Alcohol or drug abuse within three months prior to informed consent that would interfere with trial participation or any ongoing clinical condition that would jeopardize subject safety or study compliance based on investigator judgement;
* Liver disease, defined by serum levels of alanine transaminase, aspartate transaminase, or alkaline phosphatase >3 x upper limit of normal as determined during screening;
* Cardiac, lung or peripheral vascular disease or stroke;
* Pancreas, pancreatic islet cells or renal transplant recipient;
* Medical history of cancer or treatment for cancer in the last five years prior to screening;
* History of allergy or angioedema with RAAS inhibitor exposure;
* Kidney disease due primarily to another condition aside from FSGS;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
The change in Glomerular Filtration Rate (GFR) After an 8 week treatment with dapagliflozin | Before and after an 8 week treatment with dapagliflozin
  Glomerular Filtration Rate (GFR, based on plasma inulin clearance) will be measured at baseline and after 8 weeks of treatment.

SECONDARY OUTCOMES:
The change in Effective Renal Plasma Flow (ERPF) After an 8 week treatment with dapagliflozin | Before and after an 8 week treatment with dapagliflozin
  Effective Renal Plasma Flow (ERPF, based on paraaminohippurate plasma clearance) will be measured at baseline and after 8 weeks of treatment.
The change in Blood Pressure After an 8 week treatment with dapagliflozin | Before and after 8 weeks of treatment with dapagliflozin
The change in albuminuria after 8 weeks of treatment with dapagliflozin | Before and after 8 weeks of treatment with dapagliflozin
The change in urinary vasoactive mediators after 8 weeks of treatment with dapagliflozin | Before and after 8 weeks of treatment with dapagliflozin

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Physiology Laboratory, University Health Network, Toronto, Ontario, Canada